CLINICAL TRIAL: NCT05229367
Title: Mode-specific Effects of Concentric and Eccentric Isokinetic Training of Hamstring Muscle at Slow Angular Velocity on Functional Hamstrings-to-quadriceps Ratio
Brief Title: Mode Specific Effects of Isokinetic Training of Hamstring on Hamstring to Quadriceps Ratio
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King Saud University (Other)
Responsible Party: Principal Investigator, Masood Khan, Principal Investigator, King Saud University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: RRC-2021-11
Record Dates: First submitted 2022-01-27; First posted 2022-02-08 (Actual); Last update posted 2022-02-24 (Actual); Status verified 2022-02

CONDITIONS: Muscle Strength
Keywords: Isokinetic training; peak torque; acceleration time; deceleration time; time to peak torque; Hamstring-to-Quadriceps ratio

STUDY DESIGN:
Intervention Model Description: Participants were randomly divided into two groups.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Eccentric isokinetic group (Experimental): In this group, eccentric isokinetic training of hamstring muscle was performed.
  Interventions: Other: Eccentric isokinetic training
- Concentric isokinetic group (Active Comparator): In this group, concentric isokinetic training of hamstring muscle was performed.
  Interventions: Other: Concentric isokinetic training

INTERVENTIONS:
Other: Eccentric isokinetic training — Eccentric exercises of the hamstring muscles were performed with the use of an isokinetic dynamometer device.
  Arms: Eccentric isokinetic group
Other: Concentric isokinetic training — Concentric exercises of the hamstring muscles were performed with the use of an isokinetic dynamometer device.
  Arms: Concentric isokinetic group

SUMMARY:
Mode specificity of eccentric and concentric isokinetic training have been examined in previous studies but with conflicting results. The present study aimed to examine the mode-specific effects of eccentric and concentric isokinetic training of hamstring muscle at slow angular velocity on eccentric peak torque of hamstring (PTecc), concentric peak torque of quadriceps (PTcon), acceleration time of hamstring (AThams) and quadriceps (ATquad), deceleration time of hamstring (DThams) and quadriceps (DTquad), time to peak torque of hamstring (TPThams) and quadriceps (TPTquad), and functional Hamstring-to-Quadriceps ratio (PTecc/PTcon).

DETAILED DESCRIPTION:
Several studies in past have tried to examine the mode specificity of concentric and eccentric training of different muscles and at different angular velocities i.e. whether concentric training will increase the concentric strength only or both concentric and eccentric strength and whether eccentric training will increase eccentric strength only or both eccentric and concentric strength.

Since conflicting reports are available regarding mode specificity of eccentric and concentric isokinetic training therefore one study was needed that can examine the mode specificity of these training in hamstring muscles at slow angular velocity. The present study aimed to examine the mode-specific effects of six weeks of isokinetic concentric and eccentric training of the hamstring muscle at slow angular velocity on the PTecc/PTcon, AT, DT, and TPT.

ELIGIBILITY:
Inclusion Criteria:

* Healthy young males
* Age between 18 to 27
* Recreationally active who used to engage regularly in 1-5 hours of physical activity per week

Exclusion Criteria:

* Individual presently indulged in strength training of knee.
* Individuals with any kind of injury around the knee, hip, ankle, foot
* Unconsolidated fractures around the knee. • Stress fractures
* Subjects with the acute phase of trauma, which may interfere with the exercise regime
* Subjects with cardio-respiratory problems and other medical problems like diabetes, asthma, etc.
* Subjects with tendinitis and other inflammatory conditions.

Ages: 18 Years to 28 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2021-04-28 (Actual); Primary Completion 2021-09-13 (Actual); Study Completion 2021-10-14 (Actual)

PRIMARY OUTCOMES:
Functional Hamstring-to-quadriceps ratio (PTecc:PTcon) | 6 weeks
  This ratio was calculated using eccentric peak of hamstring and concentric peak torque of quadriceps muscle

SECONDARY OUTCOMES:
Acceleration time of hamstring (AThams) | 6 weeks
  Time required by hamstring muscle to reach desired velocity was noted.
Acceleration time of quadriceps | 6 weeks
  Time required by quadriceps muscle to reach desired velocity was noted.
Deceleration time of hamstring (DThams) | 6 weeks
  Time required by hamstring muscle to reach zero velocity from target velocity, was noted.
Deceleration time of quadriceps | 6 weeks
  Time required by quadriceps muscle to reach zero velocity from target velocity to, was noted.
Time to peak torque of hamstring | 6 weeks
  Time required by hamstring muscle to reach peak torque was noted.
Time to peak torque of quadriceps | 6 weeks
  Time required by quadriceps muscle to reach peak torque was noted.

CONTACTS AND LOCATIONS:
Overall Officials: Masood Khan, M.P.Th, Principal Investigator — King Saud University
Locations (1):
- King Saud University, Riyadh, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sharma KN, Quddus N, Hameed UA, Khan SA, Kumari A, Alghadir AH, Khan M. Mode-specific effects of concentric and eccentric isokinetic training of the hamstring muscle at slow angular velocity on the functional hamstrings-to-quadriceps ratio-a randomized trial. PeerJ. 2022 Sep 29;10:e13842. doi: 10.7717/peerj.13842. eCollection 2022. PMID 36196400